CLINICAL TRIAL: NCT06493890
Title: Cultural Adaptation and Validation of the Prosthesis Evaluation Questionnaire - Dutch Language Version in Lower Limb Prosthesis Users
Brief Title: Validation of the Dutch Translation of the Prosthesis Evaluation Questionnaire
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Stichting Beatrixoord Noord-Nederland (Unknown)
Responsible Party: Sponsor
Other Study IDs: MH28062024
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-12

CONDITIONS: Validation Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Validation PEQ-DLV — Validation of the Dutch Language version of the Prosthesis Evaluation Questionnaire

SUMMARY:
The aim of our research is to be able to use the questionnaire 'Prosthesis Evaluation Questionnaire' (PEQ) in Dutch. The PEQ is a validated and reliable questionnaire for research into the quality of life in adults with a lower limb prosthesis. The research consists of two phases. The first phase is the translation of the PEQ and the second phase is the validation of this questionnaire. To validate the questionnaire, we want to include 84 participants who have to complete questionnaires three times within a period of three months.

DETAILED DESCRIPTION:
The study consists of two phases. The first phase is the translation of the Prosthesis Evaluation Questionnaire (PEQ) and the second phase is the validation of this questionnaire.

Phase 1 translation PEQ: The Beaton guidelines were followed for the translation of the questionnaire. After translation and back-translation, version A of the translated PEQ was created. This version was tested on 30 adult patients with a lower leg prosthesis. Based on the feedback from the patients, the Dutch language version of the PEQ was created (PEQ-DLV).

Phase 2 validation PEQ-DLV: For the process of validation three questionnaires were used: a general survey, the PEQ-DLV and the RAND-36. The participants were approached via a large orthopedic workshop and the national patient association KorterMaarKrachtig (KMK). The aim was to include 84 lower limb prosthesis users with an unilateral amputation at ankle level or higher. At baseline (T0) patients received a digital consent form, the general survey, the PEQ-DLV and the RAND-36. Two weeks (T1) and three months (T2) after baseline, the participants who completed all questionnaires, received the PEQ-DLV again. For motivation and as a token of appreciation, participants received a compensation of 20 euros after filling in all questionnaires.During the analysis the internal consistency, floor-ceiling effects, test-retest riliability, responsiveness and contruct validity are calculated and determined.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Unilateral lower limb amputation at ankle level or higher
* Mastering Dutch language

Exclusion Criteria:

* Children
* Bilateral or foot amputations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants were approached via a large orthopedic workshop (with several locations nationwide) by mail and via the national patient association KorterMaarKrachtig (KMK) through a request on the KMK-website, Twitter, LinkedIn and Facebook-page. An information letter was provided and adult lower limb prosthesis users were able to sign up by providing their email address via a registration link. The inclusion criteria are as mentioned above. The aim was to include 84 participants. For motivation and as a token of appreciation, participants received a compensation of 20 euros.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Reliable and validated Dutch version of the PEC | T0: Baseline; T1: two weeks; T2: three months
  Cultural adaptation and validation of the Dutch translation of the Prosthesis Evaluation Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Corry K Sluis, Prof, Study Chair — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided